CLINICAL TRIAL: NCT03806855
Title: Comparisons of Health-Related Quality of Life Between Overactive Bladder-wet and -Dry Women Based on Bladder Diary
Brief Title: Health-related QoF Between OAB-wet and OAB-dry Women
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201810092RINB
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-11

CONDITIONS: Quality of Life
Keywords: Health Related Quality of Life; Overactive Bladder; Bladder Diary
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OAB-wet: The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The presence of at least one episode of urgency associated incontinence was defined to be OAB-wet.
  Interventions: Diagnostic Test: Bladder diary
- OAB-dry: The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The absence of urgency associated incontinence was defined to be OAB-dry.
  Interventions: Diagnostic Test: Bladder diary

INTERVENTIONS:
Diagnostic Test: Bladder diary — 3-day bladder diary

SUMMARY:
Overactive bladder syndrome (OAB) has a great negative impact on health-related quality of life. In literatures, few studies reported the comparisons of health related quality of life between OAB-wet and OAB-dry female patients. Thus, our aim is to compare the clinical variables and health-related quality of life between OAB-wet and OAB-dry women.

DETAILED DESCRIPTION:
Between July 2009 and January 2018, all women with OAB visiting a medical center for evaluation were reviewed. The classification of OAB-wet or OAB-dry is based on the record of the three-day bladder diary of each patient. The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The presence of at least one episode of urgency associated incontinence was defined to be OAB-wet, otherwise, OAB-dry. Besides, only female OAB patients with available King's Health Questionnaire (KHQ) data were reviewed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. More than 20-year-old
2. Female
3. Diagnosed with overactive bladder by bladder diary

Exclusion Criteria:

1. Younger than 20-year-old
2. Pregnant or planned to be pregnant

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between July 2009 and January 2018, all women older than 20-year-old with OAB visiting a medical center for evaluation were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1071 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Difference in Quality of life | Between July 2009 and January 2018
  Use questionnaire to evaluate the difference in QoF of OAB-wet and OAB-dry women

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Powell LC, Szabo SM, Walker D, Gooch K. The economic burden of overactive bladder in the United States: A systematic literature review. Neurourol Urodyn. 2018 Apr;37(4):1241-1249. doi: 10.1002/nau.23477. Epub 2018 Jan 13. PMID 29331047
- [Background] Coyne KS, Wein A, Nicholson S, Kvasz M, Chen CI, Milsom I. Economic burden of urgency urinary incontinence in the United States: a systematic review. J Manag Care Pharm. 2014 Feb;20(2):130-40. doi: 10.18553/jmcp.2014.20.2.130. PMID 24456314
- [Background] Milsom I, Coyne KS, Nicholson S, Kvasz M, Chen CI, Wein AJ. Global prevalence and economic burden of urgency urinary incontinence: a systematic review. Eur Urol. 2014 Jan;65(1):79-95. doi: 10.1016/j.eururo.2013.08.031. Epub 2013 Aug 27. PMID 24007713
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Onukwugha E, Zuckerman IH, McNally D, Coyne KS, Vats V, Mullins CD. The total economic burden of overactive bladder in the United States: a disease-specific approach. Am J Manag Care. 2009 Mar;15(4 Suppl):S90-7. PMID 19355803
- [Background] Coyne KS, Sexton CC, Bell JA, Thompson CL, Dmochowski R, Bavendam T, Chen CI, Quentin Clemens J. The prevalence of lower urinary tract symptoms (LUTS) and overactive bladder (OAB) by racial/ethnic group and age: results from OAB-POLL. Neurourol Urodyn. 2013 Mar;32(3):230-7. doi: 10.1002/nau.22295. Epub 2012 Jul 27. PMID 22847394